CLINICAL TRIAL: NCT02873286
Title: A Randomized, Single-blind, Placebo Controlled, Dose-ranging Phase II Trial in ≥ 55 Year Old Adults to Evaluate the Safety and Immunogenicity of the Recombinant MVA-BN-RSV Vaccine
Brief Title: RSV-MVA-BN Vaccine Phase II Trial in ≥ 55 Year Old Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RSV-MVA-002
Record Dates: First submitted 2016-08-09; First posted 2016-08-19 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV Vaccines; Respiratory Syncytial Virus Vaccines
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 - Single Low Dose / Booster (Experimental): First dose (Week 0): MVA-BN-RSV 1x10E8 Inf.U; Second dose (Week 4): placebo; Booster dose (Week 56): MVA-BN-RSV 1x10E8 Inf.U; (intramuscular vaccinations)
  Interventions: Biological: MVA-BN-RSV; Other: Placebo
- Group 2 - Two Low Doses (Experimental): First dose (Week 0): MVA-BN-RSV 1x10E8 Inf.U; Second dose (Week 4): MVA-BN-RSV 1x10E8 Inf.U; (intramuscular vaccinations)
  Interventions: Biological: MVA-BN-RSV
- Group 3 - Single High Dose / Booster (Experimental): First dose (Week 0): MVA-BN-RSV 5x10E8 Inf.U; Second dose (Week 4): placebo; Booster dose (Week 56): MVA-BN-RSV 5x10E8 Inf.U; (intramuscular vaccinations)
  Interventions: Biological: MVA-BN-RSV; Other: Placebo
- Group 4 - Two High Doses (Experimental): First dose (Week 0): MVA-BN-RSV 5x10E8 Inf.U; Second dose (Week 4): MVA-BN-RSV 5x10E8 Inf.U; (intramuscular vaccinations)
  Interventions: Biological: MVA-BN-RSV
- Group 5 - Placebo (Experimental): First dose (Week 0): placebo; Second dose (Week 4): placebo; (intramuscular vaccinations)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MVA-BN-RSV — MVA-mBN294B
  Arms: Group 1 - Single Low Dose / Booster; Group 2 - Two Low Doses; Group 3 - Single High Dose / Booster; Group 4 - Two High Doses
Other: Placebo — Tris Buffered Saline, sterile
  Arms: Group 1 - Single Low Dose / Booster; Group 3 - Single High Dose / Booster; Group 5 - Placebo

SUMMARY:
A total of 400 subjects will be recruited into five treatment subject groups à 80 subjects.Subject will receive two administrations 4 weeks apart which will consist of MVA-BN-RSV Dose 1, MVA-BN-RSV Dose 2 or Placebo (TBS).

86 subjects from 2 treatment groups (43 per treatment group) are supposed to receive one (booster) dose of MVA-BN-RSV vaccine approximately one year after their first vaccination. In this booster substudy, eligible subjects will receive the same dose they received during the main trial.

ELIGIBILITY:
Inclusion Criteria (Main study):

1. Male and female subjects, ≥ 55 years of age.
2. Prior to performance of any trial specific procedures, the subject has read, signed and dated an informed consent form, having been advised of the risks and benefits of the trial in a language understood by the subject, and has signed the Health Insurance Portability and Accountability Act (HIPAA) authorization form.
3. Subjects without symptomatic cardiopulmonary and/or metabolic disease. Note that subjects who have any active symptoms related to cardiac and/or pulmonary and/or metabolic disease (including e.g. uncontrolled asthma, angina pectoris, hyperglycaemia or other episodic symptoms), or who receive ongoing therapy to control current, active symptoms, are not eligible. Subjects on stable treatment (no change in ≥ 1 month) for previous and controlled symptoms or conditions are eligible. The following are examples of subjects who may bear cardiopulmonary or metabolic diagnoses but who would remain eligible:

   * Subjects on stable (no change in ≥ 1 month) therapy for findings (e.g. hypertension, hyperlipidemia) which are not associated with current symptoms or disability.
   * Subjects with type II diabetes mellitus are considered eligible as long as they are stable on oral antidiabetics and have either a documented glycated hemoglobin (HbA1c) of ≤ 8 % within three months prior to trial participation or confirmation of controlled blood glucose level must be obtained at the SCR (screening) visit by a lab test.
   * Subjects who receive short term treatment for temporary conditions.
   * Other clinically insignificant findings not deemed to be associated with increased risk for respiratory viral infections as determined by the investigator.
4. Able to comply with trial requirements; including access to transportation for trial visits.
5. Body mass index (BMI) ≥ 18.5 and ≤ 39.9

   BMI formula for pounds and inches:

   BMI = (bodyweight in pounds) * 703 (bodyheight in inches)2
6. Women of childbearing potential (WOCBP) must have used an acceptable method of contraception for at least 30 days prior to the first vaccination, must agree to use an acceptable method of contraception (as defined in Section 8.2.11) during the trial, and must avoid becoming pregnant for at least 28 days after the last vaccination. WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to each vaccination
7. Not clinically significant laboratory values as defined in the protocol, excluding any Grade ≥ 3 toxicity.
8. Negative human immunodeficiency virus antibody test (anti-HIV), negative hepatitis B surface antigen (HBsAG) and negative antibody test to hepatitis C virus.
9. Electrocardiogram (ECG) without clinically significant acute findings (e.g. findings suggestive of current ischemia, ventricular arrhythmias, congestive heart failure and ventricular hypertrophy).

Exclusion Criteria (Main Study):

1. Pregnant or breast-feeding women.
2. Uncontrolled serious infection, i.e. not responding to antimicrobial therapy.
3. History or current clinical manifestation of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject or would limit the subject's ability to complete the trial.

   * History of cerebrovascular disorders, including stroke. Patients with history of transient ischaemic attack (TIA) ≥ 1 year prior to trial participation remain eligible.
   * History of myocardial infarction within ≤ 1 year prior to trial participation, current clinical manifestation of angina pectoris, current clinical manifestation of congestive heart failure ≥ New York Heart Association (NYHA) Grade II, uncontrolled high blood pressure defined as systolic blood pressure ≥ 150 mmHg and/or diastolic ≥ 100 mmHg within the last 2 months.
4. History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement are not excluded. Persons with rheumatoid arthritis not requiring immunomodulatory and/or immunosuppressant treatment are not excluded.
5. Known or suspected impairment of immunologic functions including, but not limited to chronic inflammatory bowel disorders, diabetes mellitus type I.
6. History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision at least 6 months ago that is considered to have achieved cure. Subjects with history of skin cancer should not be vaccinated at the previous tumor site.
7. Clinically significant mental disorder, not adequately controlled by medical treatment.
8. Active or recent (within the time period of six months before trial participation) history of chronic alcohol abuse and/or intravenous and/or nasal drug abuse.
9. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. tris(hydroxymethyl)-amino methane, chicken embryo fibroblast proteins, gentamycin.
10. Known allergy to eggs or aminoglycosides.
11. History of anaphylaxis or severe allergic reaction to any vaccine.
12. Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to or after trial vaccination.
13. Having received any vaccinations or planned vaccinations with an inactivated vaccine within 14 days prior to or after trial vaccination.
14. Chronic systemic administration (defined as more than 14 days) of > 5 mg prednisone (or equivalent)/day or any other immune-modifying drugs during a period starting from three months prior to first administration of the trial vaccination and ending at the last visit of the active trial phase. The use of topical, inhaled, ophthalmic and nasal glucocorticoids is permitted.
15. Administration or planned administration of immunoglobulins and/or any blood products during a period starting from three months prior to first administration of the trial vaccination and ending at the last visit of the active trial phase.
16. Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the first trial vaccination, or planned administration of such a drug between participation in the trial and until 4 weeks after last trial vaccination.
17. Previous or planned vaccination with a RSV vaccine/vaccine candidate.
18. Clinical trial personnel working on the current trial.

Inclusion Criteria (Substudy):

1. Prior to performance of any booster substudy specific procedures, the subject has read, signed and dated an informed consent form, having been advised of the risks and benefits of the trial in a language understood by the subject.
2. Subject has completed all vaccinations of the main trial according to protocol.

Exclusion Criteria (Substudy):

1. Any condition that, in the opinion of the investigator, makes it unsafe for the subject to receive a further vaccination.
2. Pregnancy.
3. An anaphylactic reaction following the administration of any vaccine(s).
4. Clinical need for concomitant or ancillary therapy not permitted in the trial as outlined in Protocol Section 8.2.2.
5. Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to or after booster vaccination.
6. Having received any vaccinations or planned vaccinations with an inactivated vaccine within 14 days prior to or after booster vaccination.
7. Chronic systemic administration (defined as more than 14 days) of > 5 mg prednisone (or equivalent)/day or any other immune-modifying drugs during a period starting from 3 months prior to administration of the booster vaccine and ending at the last visit of the booster active trial phase. The use of topical, inhaled, ophthalmic and nasal glucocorticoids is permitted.
8. Administration or planned administration of immunoglobulins and/or any blood products during a period starting from 3 months prior to administration of the booster vaccine and ending at the last visit of the booster active trial phase.
9. Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the booster vaccination, or planned administration of such a drug during participation in the booster substudy and until 4 weeks after booster vaccination.
10. Subject's request to discontinue
11. Subject's refusal to receive booster vaccination.
12. Subject unwilling or unable to comply with trial requirements. Any reason that, in the opinion of the investigator contradicts administration of the booster vaccination or otherwise requires early discontinuation of a subject.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lawrence, MD, Principal Investigator — Washington University School of Medicine
Locations (12):
- United States (12):
  - Paradigm Research, Redding, California
  - Optimal Research, San Diego, California
  - Compass Research, The Villages, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Optimal Research, Peoria, Illinois
  - Optimal Research, Rockville, Maryland
  - Washington University in St. Louis, School of Medicine, St Louis, Missouri
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research Associates, Endwell, New York
  - Rapid Medical Research, Cleveland, Ohio
  - Ventavia Research Group, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jordan E, Lawrence SJ, Meyer TPH, Schmidt D, Schultz S, Mueller J, Stroukova D, Koenen B, Gruenert R, Silbernagl G, Vidojkovic S, Chen LM, Weidenthaler H, Samy N, Chaplin P. Broad Antibody and Cellular Immune Response From a Phase 2 Clinical Trial With a Novel Multivalent Poxvirus-Based Respiratory Syncytial Virus Vaccine. J Infect Dis. 2021 Mar 29;223(6):1062-1072. doi: 10.1093/infdis/jiaa460. PMID 32726422

RESULTS

PARTICIPANT FLOW:
Period: Main Study
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Started (Received first vaccination) | 78 | 89 | 80 | 90 | 83
Completed (Completed active trial phase) | 76 | 84 | 78 | 89 | 81
Not Completed | 2 | 5 | 2 | 1 | 2
Period: Booster Substudy
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Started (Entered substudy and received booster vaccination) | 43 | 0 | 45 | 0 | 0
Completed (Completed substudy active trial phase) | 43 | 0 | 45 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo | Total
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.09) | 64.8 (7.78) | 65.3 (7.18) | 65.0 (7.93) | 65.6 (7.20) | 65.2 (7.62)
Age, Customized [Count of Participants; unit: Participants]
  55 to 69 years | 53 | 61 | 56 | 63 | 56 | 289
  >=70 years | 25 | 28 | 24 | 27 | 27 | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 56 | 49 | 59 | 48 | 259
  Male | 31 | 33 | 31 | 31 | 35 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 1 | 4 | 1 | 16
  Not Hispanic or Latino | 75 | 82 | 79 | 86 | 82 | 404
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 0 | 2
  Black or African American | 9 | 15 | 14 | 21 | 11 | 70
  White | 69 | 69 | 66 | 69 | 71 | 344
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 78 | 89 | 80 | 90 | 83 | 420

OUTCOME MEASURES:

1. Primary Outcome: PRNT (Subtype A) GMT
Description: Geometric Mean Titers (GMTs) based on RSV-specific Plaque Reduction Neutralization Test (PRNT; against subtype A). Titers below the detection limit (DL) are included with a value of '10' (i.e. 1/2 DL)
Time Frame: Week 6 (Main Study) i.e., 2 weeks following the second vaccination
Population: Full Analysis Set i.e. all participants who received at least one vaccination in the main study. Calculations based on participants with data available for this outcome.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
Titer | 300.5 [251.7 to 358.6] | 278.9 [239.2 to 325.2] | 311.9 [261.7 to 371.7] | 373.3 [320.9 to 434.2] | 229.3 [195.2 to 269.4]

2. Secondary Outcome: PRNT (Subtype A) GMT
Description: Geometric Mean Titers (GMTs) based on RSV-specific Plaque Reduction Neutralization Test (PRNT; against subtype A). Individual peak is defined as the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Titers below the detection limit (DL) are included with a value of '10' (i.e. 1/2 DL)
Time Frame: within 108 weeks
Population: Full Analysis Set i.e. all participants who received at least one vaccination in the main study. A subset of participants from groups 1 and 3 entered the booster substudy.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Titer
  Week 0 (Main Study) | 256.4 [214.2 to 307.0] | 208.0 [180.0 to 240.3] | 234.9 [200.4 to 275.3] | 276.4 [235.9 to 323.9] | 251.7 [213.7 to 296.6]
  Week 2 (Main Study): number analyzed (Participants) | 78 | 87 | 79 | 90 | 82
  Week 2 (Main Study) | 316.7 [266.3 to 376.6] | 259.8 [222.5 to 303.4] | 356.9 [298.8 to 426.4] | 398.8 [340.8 to 466.6] | 235.0 [202.1 to 273.2]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 84 | 78 | 90 | 82
  Week 4 (Main Study) | 307.5 [259.0 to 365.2] | 258.2 [218.6 to 304.9] | 342.5 [287.5 to 408.1] | 347.7 [296.9 to 407.2] | 252.7 [214.2 to 298.0]
  Week 6 (Main Study): number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
  Week 6 (Main Study) | 300.5 [251.7 to 358.6] | 278.9 [239.2 to 325.2] | 311.9 [261.7 to 371.7] | 373.3 [320.9 to 434.2] | 229.3 [195.2 to 269.4]
  Week 8 (Main Study): number analyzed (Participants) | 77 | 85 | 79 | 89 | 81
  Week 8 (Main Study) | 292.0 [246.6 to 345.7] | 263.9 [226.9 to 306.9] | 304.0 [251.8 to 367.1] | 370.9 [316.3 to 434.9] | 231.5 [197.4 to 271.6]
  Individual Peak (Main Study): number analyzed (Participants) | 78 | 88 | 80 | 90 | 82
  Individual Peak (Main Study) | 381.7 [321.0 to 453.8] | 334.8 [287.0 to 390.6] | 450.1 [371.5 to 545.4] | 483.7 [412.5 to 567.2] | 309.9 [267.7 to 358.7]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 77 | 84 | 77 | 89 | 81
  Week 16 (Follow-Up 1) | 288.7 [236.5 to 352.4] | 261.3 [222.9 to 306.4] | 275.5 [231.1 to 328.6] | 336.5 [285.5 to 396.7] | 242.9 [204.9 to 287.8]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 75 | 83 | 76 | 88 | 82
  Week 30 (Follow-Up 2) | 244.0 [202.6 to 293.7] | 205.4 [175.5 to 240.5] | 228.2 [193.8 to 268.5] | 266.7 [228.6 to 311.1] | 202.2 [172.4 to 237.1]
  Week 56 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 56 (Booster Substudy) | 285.6 [228.4 to 357.1] |  | 264.2 [218.9 to 318.9] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 58 (Booster Substudy) | 351.9 [275.4 to 449.7] |  | 286.0 [236.0 to 346.7] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 60 (Booster Substudy) | 402.1 [323.9 to 499.2] |  | 341.2 [281.0 to 414.3] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Individual Peak (Booster Substudy) | 424.3 [339.6 to 530.3] |  | 358.6 [296.9 to 433.1] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 287.9 [231.3 to 358.4] |  | 235.9 [195.6 to 284.5] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 405.8 [312.0 to 527.7] |  | 333.9 [271.4 to 411.0] |  |
  Week 108 (Booster Follow-Up 3): number analyzed (Participants) | 43 | 0 | 44 | 0 | 0
  Week 108 (Booster Follow-Up 3) | 296.2 [235.1 to 373.1] |  | 258.1 [210.6 to 316.4] |  |

3. Secondary Outcome: Percentage of Participants With Response by PRNT (Subtype A)
Description: Response rate based on RSV-specific Plaque Reduction Neutralization Test (PRNT; against subtype A). Response is defined as the appearance of antibody titers ≥ detection limit (20) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Individual peak response rate is based on the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Percentages based on number of subjects with data available.
Time Frame: within 108 weeks
Population: Full Analysis Set i.e. all participants who received at least one vaccination in the main study. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline. A subset of participants from groups 1 and 3 entered the booster substudy.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 88 | 79 | 90 | 82
percentage of subjects
  Week 2 (Main Study): number analyzed (Participants) | 78 | 87 | 79 | 90 | 82
  Week 2 (Main Study) | 10.3 [4.5 to 19.2] | 9.2 [4.1 to 17.3] | 27.8 [18.3 to 39.1] | 23.3 [15.1 to 33.4] | 3.7 [0.8 to 10.3]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 84 | 78 | 90 | 82
  Week 4 (Main Study) | 13.3 [6.6 to 23.2] | 11.9 [5.9 to 20.8] | 25.6 [16.4 to 36.8] | 8.9 [3.9 to 16.8] | 1.2 [0.0 to 6.6]
  Week 6 (Main Study): number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
  Week 6 (Main Study) | 9.2 [3.8 to 18.1] | 15.5 [8.5 to 25.0] | 19.2 [11.2 to 29.7] | 15.6 [8.8 to 24.7] | 4.9 [1.4 to 12.2]
  Week 8 (Main Study): number analyzed (Participants) | 77 | 85 | 79 | 89 | 81
  Week 8 (Main Study) | 7.8 [2.9 to 16.2] | 10.6 [5.0 to 19.2] | 15.2 [8.1 to 25.0] | 14.6 [8.0 to 23.7] | 1.2 [0.0 to 6.7]
  Individual Peak (Main Study) | 23.1 [14.3 to 34.0] | 25.0 [16.4 to 35.4] | 41.3 [30.4 to 52.8] | 34.4 [24.7 to 45.2] | 7.3 [2.7 to 15.2]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 77 | 84 | 77 | 89 | 81
  Week 16 (Follow-Up 1) | 9.1 [3.7 to 17.8] | 8.3 [3.4 to 16.4] | 10.4 [4.6 to 19.4] | 10.1 [4.7 to 18.3] | 4.9 [1.4 to 12.2]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 75 | 83 | 76 | 88 | 82
  Week 30 (Follow-Up 2) | 1.3 [0.0 to 7.2] | 7.2 [2.7 to 15.1] | 3.9 [0.8 to 11.1] | 2.3 [0.3 to 8.0] | 3.7 [0.8 to 10.3]
  Week 58 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 58 (Booster Substudy) | 17.1 [7.2 to 32.1] |  | 4.4 [0.5 to 15.1] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 60 (Booster Substudy) | 19.5 [8.8 to 34.9] |  | 11.1 [3.7 to 24.1] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Individual Peak (Booster Substudy) | 22.0 [10.6 to 37.6] |  | 15.6 [6.5 to 29.5] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 2.4 [0.1 to 12.9] |  | 0.0 [0.0 to 7.9] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 22.0 [10.6 to 37.6] |  | 13.3 [5.1 to 26.8] |  |
  Week 108 (Booster Follow-Up 3): number analyzed (Participants) | 41 | 0 | 44 | 0 | 0
  Week 108 (Booster Follow-Up 3) | 2.4 [0.1 to 12.9] |  | 4.5 [0.6 to 15.5] |  |

4. Secondary Outcome: PRNT (Subtype B) GMT
Description: Geometric Mean Titers (GMTs) based on RSV-specific Plaque Reduction Neutralization Test (PRNT; against subtype B). Individual peak is defined as the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Titers below the detection limit (DL) are included with a value of '10' (i.e. 1/2 DL)
Time Frame: within 108 weeks
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Titer
  Week 0 (Main Study) | 424.3 [332.0 to 542.2] | 364.9 [285.6 to 466.2] | 426.9 [331.7 to 549.4] | 498.6 [395.6 to 628.5] | 477.5 [361.3 to 630.9]
  Week 2 (Main Study): number analyzed (Participants) | 78 | 87 | 79 | 90 | 82
  Week 2 (Main Study) | 517.7 [407.4 to 657.9] | 464.5 [363.7 to 593.3] | 688.6 [528.6 to 896.9] | 638.2 [510.9 to 797.3] | 441.4 [331.6 to 587.6]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 84 | 78 | 90 | 82
  Week 4 (Main Study) | 485.8 [385.9 to 611.4] | 458.8 [355.3 to 592.6] | 635.9 [490.6 to 824.1] | 570.0 [453.6 to 716.3] | 431.5 [325.3 to 572.4]
  Week 6 (Main Study): number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
  Week 6 (Main Study) | 506.1 [395.0 to 648.4] | 507.4 [396.4 to 649.6] | 615.1 [468.9 to 806.8] | 674.3 [544.9 to 834.4] | 454.0 [340.7 to 605.0]
  Week 8 (Main Study): number analyzed (Participants) | 77 | 85 | 79 | 89 | 81
  Week 8 (Main Study) | 509.0 [398.4 to 650.5] | 483.5 [379.5 to 615.9] | 670.1 [505.4 to 888.5] | 610.2 [492.5 to 756.0] | 465.3 [351.8 to 615.5]
  Individual Peak (Main Study): number analyzed (Participants) | 78 | 88 | 80 | 90 | 82
  Individual Peak (Main Study) | 672.2 [531.5 to 850.2] | 639.7 [503.1 to 813.3] | 932.3 [702.7 to 1236.9] | 858.0 [689.2 to 1068.0] | 614.6 [462.0 to 817.8]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 77 | 84 | 77 | 89 | 81
  Week 16 (Follow-Up 1) | 577.8 [457.1 to 730.5] | 505.7 [403.4 to 634.0] | 639.0 [499.4 to 817.7] | 635.6 [517.1 to 781.1] | 515.6 [394.3 to 674.3]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 75 | 83 | 76 | 88 | 82
  Week 30 (Follow-Up 2) | 570.6 [453.7 to 717.6] | 458.1 [361.9 to 579.8] | 606.1 [479.9 to 765.3] | 583.2 [471.2 to 721.9] | 518.1 [398.7 to 673.3]
  Week 56 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 56 (Booster Substudy) | 561.0 [395.7 to 795.3] |  | 584.5 [423.4 to 806.9] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 58 (Booster Substudy) | 894.1 [656.2 to 1218.2] |  | 954.8 [702.8 to 1297.0] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 60 (Booster Substudy) | 761.7 [561.4 to 1033.4] |  | 804.2 [585.9 to 1103.9] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Individual Peak (Booster Substudy) | 992.5 [730.1 to 1349.2] |  | 1031.2 [755.2 to 1407.9] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 632.2 [470.4 to 849.5] |  | 686.7 [509.1 to 926.4] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 759.0 [561.3 to 1026.5] |  | 782.3 [581.8 to 1051.9] |  |
  Week 108 (Booster Follow-Up 3): number analyzed (Participants) | 43 | 0 | 44 | 0 | 0
  Week 108 (Booster Follow-Up 3) | 599.7 [448.8 to 801.3] |  | 669.4 [493.7 to 907.6] |  |

5. Secondary Outcome: Percentage of Participants With Response by PRNT (Subtype B)
Description: Response rate based on RSV-specific Plaque Reduction Neutralization Test (PRNT; against subtype B). Response is defined as the appearance of antibody titers ≥ detection limit (20) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Individual peak response rate is based on the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Percentages based on number of subjects with data available.
Time Frame: within 108 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 88 | 79 | 90 | 82
percentage of subjects
  Week 2 (Main Study): number analyzed (Participants) | 78 | 87 | 79 | 90 | 82
  Week 2 (Main Study) | 12.8 [6.3 to 22.3] | 18.4 [10.9 to 28.1] | 26.6 [17.3 to 37.7] | 14.4 [7.9 to 23.4] | 2.4 [0.3 to 8.5]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 84 | 78 | 90 | 82
  Week 4 (Main Study) | 9.3 [3.8 to 18.3] | 14.3 [7.6 to 23.6] | 29.5 [19.7 to 40.9] | 11.1 [5.5 to 19.5] | 2.4 [0.3 to 8.5]
  Week 6 (Main Study): number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
  Week 6 (Main Study) | 10.5 [4.7 to 19.7] | 21.4 [13.2 to 31.7] | 24.4 [15.3 to 35.4] | 21.1 [13.2 to 31.0] | 4.9 [1.4 to 12.2]
  Week 8 (Main Study): number analyzed (Participants) | 77 | 85 | 79 | 89 | 81
  Week 8 (Main Study) | 15.6 [8.3 to 25.6] | 11.8 [5.8 to 20.6] | 26.6 [17.3 to 37.7] | 14.6 [8.0 to 23.7] | 2.5 [0.3 to 8.6]
  Individual Peak (Main Study) | 25.6 [16.4 to 36.8] | 34.1 [24.3 to 45.0] | 45.0 [33.8 to 56.5] | 34.4 [24.7 to 45.2] | 9.8 [4.3 to 18.3]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 77 | 84 | 77 | 89 | 81
  Week 16 (Follow-Up 1) | 11.7 [5.5 to 21.0] | 20.2 [12.3 to 30.4] | 22.1 [13.4 to 33.0] | 13.5 [7.2 to 22.4] | 7.4 [2.8 to 15.4]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 75 | 83 | 76 | 88 | 82
  Week 30 (Follow-Up 2) | 20.0 [11.6 to 30.8] | 13.3 [6.8 to 22.5] | 21.1 [12.5 to 31.9] | 11.4 [5.6 to 19.9] | 11.0 [5.1 to 19.8]
  Week 58 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 58 (Booster Substudy) | 39.0 [24.2 to 55.5] |  | 33.3 [20.0 to 49.0] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 60 (Booster Substudy) | 17.1 [7.2 to 32.1] |  | 20.0 [9.6 to 34.6] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Individual Peak (Booster Substudy) | 39.0 [24.2 to 55.5] |  | 35.6 [21.9 to 51.2] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 14.6 [5.6 to 29.2] |  | 11.1 [3.7 to 24.1] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 19.5 [8.8 to 34.9] |  | 17.8 [8.0 to 32.1] |  |
  Week 108 (Booster Follow-Up 3): number analyzed (Participants) | 41 | 0 | 44 | 0 | 0
  Week 108 (Booster Follow-Up 3) | 4.9 [0.6 to 16.5] |  | 9.1 [2.5 to 21.7] |  |

6. Secondary Outcome: ELISA (IgG) GMT
Description: Geometric Mean Titers (GMTs) based on RSV-specific Immunoglobulin G (IgG) Enzyme-linked Immunosorbent Assay (ELISA). Individual peak is defined as the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Titers below the detection limit (DL) are included with a value of '31.5' (i.e. 1/2 DL)
Time Frame: within 108 weeks
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Titer
  Week 0 (Main Study) | 1578.4 [1394.0 to 1787.3] | 1488.6 [1322.4 to 1675.8] | 1636.1 [1421.9 to 1882.6] | 1819.5 [1595.2 to 2075.2] | 1672.2 [1480.7 to 1888.4]
  Week 2 (Main Study): number analyzed (Participants) | 78 | 87 | 79 | 90 | 82
  Week 2 (Main Study) | 2506.9 [2221.3 to 2829.3] | 2460.0 [2172.9 to 2785.0] | 3773.6 [3212.8 to 4432.4] | 3639.5 [3212.7 to 4122.9] | 1674.3 [1486.8 to 1885.5]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 84 | 78 | 90 | 82
  Week 4 (Main Study) | 2599.9 [2299.0 to 2940.2] | 2559.9 [2233.4 to 2934.2] | 3884.6 [3336.2 to 4523.2] | 3697.0 [3257.6 to 4195.7] | 1747.3 [1550.1 to 1969.6]
  Week 6 (Main Study): number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
  Week 6 (Main Study) | 2671.0 [2365.5 to 3015.9] | 2964.1 [2601.4 to 3377.2] | 3864.3 [3348.1 to 4460.2] | 4270.0 [3753.4 to 4857.7] | 1766.6 [1536.0 to 2031.8]
  Week 8 (Main Study): number analyzed (Participants) | 77 | 85 | 79 | 89 | 81
  Week 8 (Main Study) | 2653.4 [2309.5 to 3048.5] | 2960.1 [2592.8 to 3379.4] | 3773.6 [3278.4 to 4343.6] | 4283.2 [3790.3 to 4840.2] | 1844.6 [1603.1 to 2122.5]
  Individual Peak (Main Study): number analyzed (Participants) | 78 | 88 | 80 | 90 | 82
  Individual Peak (Main Study) | 3266.2 [2878.5 to 3706.1] | 3412.2 [3001.8 to 3878.8] | 4824.0 [4161.9 to 5591.4] | 5061.4 [4493.0 to 5701.8] | 2207.2 [1926.4 to 2528.8]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 77 | 84 | 77 | 89 | 81
  Week 16 (Follow-Up 1) | 2833.4 [2489.8 to 3224.3] | 2965.0 [2609.3 to 3369.3] | 3294.5 [2906.5 to 3734.2] | 3950.8 [3519.2 to 4435.3] | 2117.1 [1815.8 to 2468.3]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 75 | 83 | 76 | 88 | 82
  Week 30 (Follow-Up 2) | 2162.3 [1885.3 to 2480.2] | 2107.5 [1825.7 to 2432.7] | 2796.5 [2416.3 to 3236.6] | 3023.4 [2682.7 to 3407.3] | 1777.6 [1513.1 to 2088.4]
  Week 56 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 56 (Booster Substudy) | 2501.8 [2145.8 to 2916.8] |  | 2816.4 [2406.9 to 3295.5] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 58 (Booster Substudy) | 3878.2 [3263.2 to 4609.1] |  | 4261.7 [3532.7 to 5141.1] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 60 (Booster Substudy) | 4139.6 [3466.7 to 4943.2] |  | 4368.3 [3622.1 to 5268.2] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Individual Peak (Booster Substudy) | 4445.5 [3730.1 to 5298.1] |  | 4788.9 [3970.0 to 5776.8] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 3031.5 [2489.7 to 3691.2] |  | 3250.5 [2652.3 to 3983.6] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 2568.9 [2169.2 to 3042.3] |  | 2754.0 [2335.0 to 3248.1] |  |
  Week 108 (Booster Follow-Up 3): number analyzed (Participants) | 43 | 0 | 44 | 0 | 0
  Week 108 (Booster Follow-Up 3) | 2083.1 [1761.6 to 2463.4] |  | 2260.0 [1893.7 to 2697.0] |  |

7. Secondary Outcome: Percentage of Participants With Response by IgG ELISA
Description: Response rate based on RSV-specific Immunoglobulin G (IgG) Enzyme-linked Immunosorbent Assay (ELISA). Response is defined as the appearance of antibody titers ≥ detection limit (63) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Individual peak response rate is based on the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Percentages based on number of subjects with data available.
Time Frame: within 108 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 88 | 79 | 90 | 82
percentage of subjects
  Week 2 (Main Study): number analyzed (Participants) | 78 | 87 | 79 | 90 | 82
  Week 2 (Main Study) | 21.8 [13.2 to 32.6] | 19.5 [11.8 to 29.4] | 51.9 [40.4 to 63.3] | 44.4 [34.0 to 55.3] | 0.0 [0.0 to 4.4]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 84 | 78 | 90 | 82
  Week 4 (Main Study) | 24.0 [14.9 to 35.3] | 27.4 [18.2 to 38.2] | 60.3 [48.5 to 71.2] | 46.7 [36.1 to 57.5] | 2.4 [0.3 to 8.5]
  Week 6 (Main Study): number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
  Week 6 (Main Study) | 28.9 [19.1 to 40.5] | 39.3 [28.8 to 50.5] | 55.1 [43.4 to 66.4] | 58.9 [48.0 to 69.2] | 2.5 [0.3 to 8.6]
  Week 8 (Main Study): number analyzed (Participants) | 77 | 85 | 79 | 89 | 81
  Week 8 (Main Study) | 29.9 [20.0 to 41.4] | 40.0 [29.5 to 51.2] | 54.4 [42.8 to 65.7] | 59.6 [48.6 to 69.8] | 1.2 [0.0 to 6.7]
  Individual Peak (Main Study) | 42.3 [31.2 to 54.0] | 53.4 [42.5 to 64.1] | 70.0 [58.7 to 79.7] | 71.1 [60.6 to 80.2] | 4.9 [1.3 to 12.0]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 77 | 84 | 77 | 89 | 81
  Week 16 (Follow-Up 1) | 29.9 [20.0 to 41.4] | 44.0 [33.2 to 55.3] | 45.5 [34.1 to 57.2] | 51.7 [40.8 to 62.4] | 7.4 [2.8 to 15.4]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 75 | 83 | 76 | 88 | 82
  Week 30 (Follow-Up 2) | 13.3 [6.6 to 23.2] | 14.5 [7.7 to 23.9] | 28.9 [19.1 to 40.5] | 26.1 [17.3 to 36.6] | 7.3 [2.7 to 15.2]
  Week 58 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 58 (Booster Substudy) | 22.0 [10.6 to 37.6] |  | 22.2 [11.2 to 37.1] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 60 (Booster Substudy) | 19.5 [8.8 to 34.9] |  | 17.8 [8.0 to 32.1] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Individual Peak (Booster Substudy) | 24.4 [12.4 to 40.3] |  | 28.9 [16.4 to 44.3] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 9.8 [2.7 to 23.1] |  | 13.3 [5.1 to 26.8] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 4.9 [0.6 to 16.5] |  | 4.4 [0.5 to 15.1] |  |
  Week 108 (Booster Follow-Up 3): number analyzed (Participants) | 41 | 0 | 44 | 0 | 0
  Week 108 (Booster Follow-Up 3) | 0.0 [0.0 to 8.6] |  | 4.5 [0.6 to 15.5] |  |

8. Secondary Outcome: ELISA (IgA) GMT
Description: Geometric Mean Titers (GMTs) based on RSV-specific Immunoglobulin A (IgA) Enzyme-linked Immunosorbent Assay (ELISA). Individual peak is defined as the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Titers below the detection limit (DL) are included with a value of '50' (i.e. 1/2 DL)
Time Frame: within 108 weeks
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Titer
  Week 0 (Main Study) | 581.7 [453.0 to 747.1] | 591.1 [475.1 to 735.3] | 776.3 [614.9 to 980.0] | 623.3 [494.9 to 785.0] | 585.4 [451.7 to 758.5]
  Week 2 (Main Study): number analyzed (Participants) | 78 | 87 | 79 | 90 | 82
  Week 2 (Main Study) | 1377.7 [1091.6 to 1738.7] | 1373.3 [1067.2 to 1767.1] | 2593.6 [2017.9 to 3333.6] | 1922.8 [1515.9 to 2439.0] | 619.8 [487.6 to 787.8]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 84 | 78 | 90 | 82
  Week 4 (Main Study) | 1061.3 [813.6 to 1384.5] | 1120.8 [858.2 to 1463.8] | 1763.0 [1370.6 to 2267.7] | 1378.1 [1091.0 to 1740.7] | 614.9 [478.3 to 790.7]
  Week 6 (Main Study): number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
  Week 6 (Main Study) | 1001.3 [778.6 to 1287.7] | 1248.3 [958.1 to 1626.4] | 1538.8 [1205.5 to 1964.1] | 1592.9 [1279.9 to 1982.4] | 608.8 [462.1 to 802.0]
  Week 8 (Main Study): number analyzed (Participants) | 77 | 85 | 79 | 89 | 81
  Week 8 (Main Study) | 887.3 [687.6 to 1145.1] | 1045.1 [808.6 to 1350.9] | 1459.2 [1137.2 to 1872.4] | 1367.3 [1071.6 to 1744.6] | 590.8 [447.9 to 779.4]
  Individual Peak (Main Study): number analyzed (Participants) | 78 | 88 | 80 | 90 | 82
  Individual Peak (Main Study) | 1511.0 [1195.9 to 1909.1] | 1696.5 [1336.9 to 2152.8] | 2795.1 [2173.6 to 3594.1] | 2331.1 [1860.6 to 2920.8] | 777.0 [601.7 to 1003.5]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 77 | 84 | 77 | 89 | 81
  Week 16 (Follow-Up 1) | 745.3 [580.6 to 956.7] | 709.8 [550.2 to 915.5] | 1001.6 [786.2 to 1276.1] | 933.2 [754.0 to 1155.1] | 573.8 [439.6 to 748.9]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 75 | 83 | 76 | 88 | 82
  Week 30 (Follow-Up 2) | 675.3 [531.3 to 858.4] | 743.5 [568.8 to 971.9] | 1089.5 [887.7 to 1337.2] | 970.3 [796.6 to 1181.8] | 676.3 [534.5 to 855.7]
  Week 56 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 56 (Booster Substudy) | 627.3 [437.3 to 899.8] |  | 719.4 [540.8 to 957.0] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 58 (Booster Substudy) | 1235.2 [864.0 to 1766.0] |  | 1480.5 [1153.1 to 1900.8] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 60 (Booster Substudy) | 941.3 [658.9 to 1344.7] |  | 1099.0 [829.3 to 1456.4] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Individual Peak (Booster Substudy) | 1261.3 [887.5 to 1792.5] |  | 1511.0 [1175.0 to 1943.0] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 734.4 [513.4 to 1050.5] |  | 853.3 [629.1 to 1157.3] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 711.0 [517.8 to 976.2] |  | 838.1 [649.2 to 1081.9] |  |
  Week 108 (Booster Follow-Up 3): number analyzed (Participants) | 43 | 0 | 44 | 0 | 0
  Week 108 (Booster Follow-Up 3) | 619.1 [448.7 to 854.3] |  | 716.7 [542.0 to 947.7] |  |

9. Secondary Outcome: Percentage of Participants With Response by IgA ELISA
Description: Response rate based on RSV-specific Immunoglobulin A (IgA) Enzyme-linked Immunosorbent Assay (ELISA). Response is defined as the appearance of antibody titers ≥ detection limit (100) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Individual peak response rate is based on the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Percentages based on number of subjects with data available.
Time Frame: within 108 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 88 | 79 | 90 | 82
percentage of subjects
  Week 2 (Main Study): number analyzed (Participants) | 78 | 87 | 79 | 90 | 82
  Week 2 (Main Study) | 50.0 [38.5 to 61.5] | 51.7 [40.8 to 62.6] | 68.4 [56.9 to 78.4] | 70.0 [59.4 to 79.2] | 7.3 [2.7 to 15.2]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 84 | 78 | 90 | 82
  Week 4 (Main Study) | 32.0 [21.7 to 43.8] | 36.9 [26.6 to 48.1] | 48.7 [37.2 to 60.3] | 52.2 [41.4 to 62.9] | 7.3 [2.7 to 15.2]
  Week 6 (Main Study): number analyzed (Participants) | 76 | 84 | 78 | 90 | 81
  Week 6 (Main Study) | 28.9 [19.1 to 40.5] | 46.4 [35.5 to 57.6] | 44.9 [33.6 to 56.6] | 62.2 [51.4 to 72.2] | 3.7 [0.8 to 10.4]
  Week 8 (Main Study): number analyzed (Participants) | 77 | 85 | 79 | 89 | 81
  Week 8 (Main Study) | 24.7 [15.6 to 35.8] | 37.6 [27.4 to 48.8] | 36.7 [26.1 to 48.3] | 51.7 [40.8 to 62.4] | 4.9 [1.4 to 12.2]
  Individual Peak (Main Study) | 53.8 [42.2 to 65.2] | 69.3 [58.6 to 78.7] | 72.5 [61.4 to 81.9] | 77.8 [67.8 to 85.9] | 14.6 [7.8 to 24.2]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 77 | 84 | 77 | 89 | 81
  Week 16 (Follow-Up 1) | 14.3 [7.4 to 24.1] | 14.3 [7.6 to 23.6] | 28.6 [18.8 to 40.0] | 22.5 [14.3 to 32.6] | 8.6 [3.5 to 17.0]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 75 | 83 | 76 | 88 | 82
  Week 30 (Follow-Up 2) | 9.3 [3.8 to 18.3] | 22.9 [14.4 to 33.4] | 27.6 [18.0 to 39.1] | 30.7 [21.3 to 41.4] | 14.6 [7.8 to 24.2]
  Week 58 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 58 (Booster Substudy) | 39.0 [24.2 to 55.5] |  | 44.4 [29.6 to 60.0] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 60 (Booster Substudy) | 17.1 [7.2 to 32.1] |  | 24.4 [12.9 to 39.5] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Individual Peak (Booster Substudy) | 39.0 [24.2 to 55.5] |  | 44.4 [29.6 to 60.0] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 7.3 [1.5 to 19.9] |  | 6.7 [1.4 to 18.3] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 41 | 0 | 45 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 7.3 [1.5 to 19.9] |  | 2.2 [0.1 to 11.8] |  |
  Week 108 (Booster Follow-Up 3): number analyzed (Participants) | 41 | 0 | 44 | 0 | 0
  Week 108 (Booster Follow-Up 3) | 2.4 [0.1 to 12.9] |  | 0.0 [0.0 to 8.0] |  |

10. Secondary Outcome: ELISA (Mucosal IgA) GMT
Description: Geometric Mean Titers (GMTs) based on mucosal RSV-specific Immunoglobulin A (IgA) Enzyme-linked Immunosorbent Assay (ELISA). Individual peak is defined as the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Titers below the detection limit (DL) are included with a value of '1' (i.e. 1/2 DL)
Time Frame: within 82 weeks
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 77 | 89 | 80 | 90 | 83
Titer
  Week 0 (Main Study): number analyzed (Participants) | 76 | 88 | 79 | 88 | 79
  Week 0 (Main Study) | 12.0 [9.8 to 14.6] | 10.9 [9.4 to 12.5] | 11.9 [9.7 to 14.6] | 13.7 [11.4 to 16.6] | 12.3 [10.1 to 14.8]
  Week 2 (Main Study): number analyzed (Participants) | 75 | 84 | 77 | 90 | 80
  Week 2 (Main Study) | 14.1 [11.7 to 17.0] | 12.1 [10.3 to 14.3] | 15.7 [13.3 to 18.5] | 15.2 [12.6 to 18.3] | 12.0 [9.9 to 14.7]
  Week 4 (Main Study): number analyzed (Participants) | 75 | 80 | 75 | 88 | 80
  Week 4 (Main Study) | 13.6 [11.4 to 16.1] | 13.1 [11.2 to 15.3] | 14.1 [11.9 to 16.7] | 15.0 [12.6 to 17.8] | 12.2 [10.2 to 14.7]
  Week 6 (Main Study): number analyzed (Participants) | 73 | 80 | 74 | 87 | 77
  Week 6 (Main Study) | 13.1 [10.9 to 15.7] | 13.4 [11.3 to 15.8] | 13.2 [11.0 to 15.7] | 15.1 [12.7 to 18.1] | 12.4 [10.1 to 15.2]
  Week 8 (Main Study): number analyzed (Participants) | 76 | 80 | 76 | 86 | 78
  Week 8 (Main Study) | 13.5 [11.4 to 15.9] | 12.6 [10.9 to 14.6] | 13.1 [10.8 to 15.7] | 14.6 [12.1 to 17.5] | 11.2 [9.1 to 13.8]
  Individual Peak (Main Study): number analyzed (Participants) | 77 | 88 | 79 | 90 | 82
  Individual Peak (Main Study) | 18.6 [15.8 to 21.9] | 18.0 [15.3 to 21.1] | 20.5 [17.5 to 24.0] | 21.4 [18.0 to 25.4] | 17.3 [14.4 to 20.8]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 74 | 83 | 76 | 86 | 80
  Week 16 (Follow-Up 1) | 13.0 [10.7 to 15.8] | 11.9 [10.0 to 14.0] | 13.2 [10.9 to 16.2] | 13.0 [10.7 to 15.8] | 11.7 [9.7 to 14.1]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 73 | 81 | 76 | 85 | 79
  Week 30 (Follow-Up 2) | 13.1 [11.2 to 15.3] | 12.1 [10.3 to 14.2] | 13.4 [11.0 to 16.2] | 13.6 [11.4 to 16.2] | 13.1 [10.6 to 16.1]
  Week 56 (Booster Substudy): number analyzed (Participants) | 42 | 0 | 42 | 0 | 0
  Week 56 (Booster Substudy) | 15.6 [12.8 to 19.0] |  | 11.9 [9.5 to 14.9] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 43 | 0 | 0
  Week 58 (Booster Substudy) | 15.0 [12.0 to 18.8] |  | 14.6 [11.6 to 18.3] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 41 | 0 | 0
  Week 60 (Booster Substudy) | 16.4 [13.4 to 20.1] |  | 13.8 [11.1 to 17.2] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 42 | 0 | 43 | 0 | 0
  Individual Peak (Booster Substudy) | 18.2 [15.1 to 21.9] |  | 16.5 [13.4 to 20.4] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 41 | 0 | 43 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 16.9 [13.8 to 20.6] |  | 13.3 [10.5 to 16.8] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 40 | 0 | 43 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 12.7 [9.6 to 16.6] |  | 8.4 [6.5 to 11.0] |  |

11. Secondary Outcome: Percentage of Participants With Response by Mucosal IgA ELISA
Description: Response rate based on mucosal RSV-specific Immunoglobulin A (IgA) Enzyme-linked Immunosorbent Assay (ELISA). Response is defined as the appearance of antibody titers ≥ detection limit (2) for initially negative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Individual peak response rate is based on the maximum post-Baseline antibody titer up to the end of the respective active trial phase i.e., within 8 weeks for the main study and within 4 weeks for the booster substudy. Percentages based on number of subjects with data available.
Time Frame: within 82 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 76 | 87 | 78 | 88 | 78
percentage of subjects
  Week 2 (Main Study): number analyzed (Participants) | 74 | 83 | 76 | 88 | 78
  Week 2 (Main Study) | 12.2 [5.7 to 21.8] | 14.5 [7.7 to 23.9] | 22.4 [13.6 to 33.4] | 12.5 [6.4 to 21.3] | 5.1 [1.4 to 12.6]
  Week 4 (Main Study): number analyzed (Participants) | 74 | 79 | 74 | 86 | 77
  Week 4 (Main Study) | 14.9 [7.7 to 25.0] | 12.7 [6.2 to 22.0] | 13.5 [6.7 to 23.5] | 14.0 [7.4 to 23.1] | 10.4 [4.6 to 19.4]
  Week 6 (Main Study): number analyzed (Participants) | 72 | 79 | 74 | 85 | 74
  Week 6 (Main Study) | 12.5 [5.9 to 22.4] | 17.7 [10.0 to 27.9] | 17.6 [9.7 to 28.2] | 16.5 [9.3 to 26.1] | 8.1 [3.0 to 16.8]
  Week 8 (Main Study): number analyzed (Participants) | 75 | 79 | 75 | 84 | 75
  Week 8 (Main Study) | 13.3 [6.6 to 23.2] | 16.5 [9.1 to 26.5] | 20.0 [11.6 to 30.8] | 11.9 [5.9 to 20.8] | 6.7 [2.2 to 14.9]
  Individual Peak (Main Study) | 25.0 [15.8 to 36.3] | 34.5 [24.6 to 45.4] | 33.3 [23.1 to 44.9] | 28.4 [19.3 to 39.0] | 17.9 [10.2 to 28.3]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 73 | 82 | 75 | 84 | 78
  Week 16 (Follow-Up 1) | 12.3 [5.8 to 22.1] | 15.9 [8.7 to 25.6] | 18.7 [10.6 to 29.3] | 11.9 [5.9 to 20.8] | 7.7 [2.9 to 16.0]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 72 | 80 | 75 | 84 | 78
  Week 30 (Follow-Up 2) | 12.5 [5.9 to 22.4] | 12.5 [6.2 to 21.8] | 20.0 [11.6 to 30.8] | 10.7 [5.0 to 19.4] | 11.5 [5.4 to 20.8]
  Week 58 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 42 | 0 | 0
  Week 58 (Booster Substudy) | 12.2 [4.1 to 26.2] |  | 7.1 [1.5 to 19.5] |  |
  Week 60 (Booster Substudy): number analyzed (Participants) | 41 | 0 | 40 | 0 | 0
  Week 60 (Booster Substudy) | 12.2 [4.1 to 26.2] |  | 2.5 [0.1 to 13.2] |  |
  Individual Peak (Booster Substudy): number analyzed (Participants) | 42 | 0 | 42 | 0 | 0
  Individual Peak (Booster Substudy) | 14.3 [5.4 to 28.5] |  | 9.5 [2.7 to 22.6] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 41 | 0 | 42 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 7.3 [1.5 to 19.9] |  | 9.5 [2.7 to 22.6] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 40 | 0 | 42 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 15.0 [5.7 to 29.8] |  | 0.0 [0.0 to 8.4] |  |

12. Secondary Outcome: ELISPOT (IFN-g, Peptide Pool: F) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool F. Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: Immunogenicity Analysis Set i.e. all participants who received at least one vaccination in the main study and were assigned to the subgroup for Peripheral Blood Mononuclear Cells (PBMC) collection. A subset of participants from groups 1 and 3 entered the booster substudy.
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 283.2 [210.1 to 381.7] | 141.3 [88.9 to 224.6] | 142.6 [85.4 to 238.3] | 245.8 [162.2 to 372.2] | 138.9 [83.8 to 230.2]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 683.3 [511.3 to 913.2] | 662.9 [475.7 to 923.8] | 940.4 [719.8 to 1228.7] | 810.2 [592.9 to 1107.1] | 117.1 [70.6 to 194.1]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 589.5 [447.2 to 777.3] | 384.9 [218.7 to 677.2] | 591.0 [438.7 to 796.2] | 598.2 [446.1 to 802.1] | 144.3 [94.6 to 220.1]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 420.1 [291.0 to 606.4] | 353.4 [253.1 to 493.5] | 496.4 [353.1 to 697.7] | 608.6 [459.2 to 806.5] | 140.9 [84.0 to 236.3]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 392.5 [258.6 to 595.8] | 348.9 [218.3 to 557.7] | 502.8 [346.8 to 728.9] | 553.1 [428.5 to 713.9] | 122.9 [76.3 to 197.9]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 282.6 [190.6 to 418.9] |  | 378.8 [185.6 to 773.4] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 628.7 [432.7 to 913.6] |  | 566.2 [349.4 to 917.5] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 514.4 [365.5 to 723.9] |  | 539.7 [325.5 to 894.7] |  |

13. Secondary Outcome: ELISPOT (IFN-g, Peptide Pool: G(A)) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool G(A). Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 124.2 [75.3 to 205.0] | 70.2 [44.6 to 110.4] | 66.2 [43.0 to 101.9] | 150.7 [101.1 to 224.6] | 88.1 [54.5 to 142.5]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 517.9 [369.1 to 726.8] | 370.9 [219.2 to 627.6] | 564.7 [395.2 to 807.1] | 659.7 [436.3 to 997.5] | 68.2 [40.9 to 113.8]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 369.3 [245.8 to 555.0] | 190.5 [100.6 to 360.7] | 290.0 [169.5 to 496.1] | 432.7 [337.0 to 555.5] | 71.2 [41.3 to 122.7]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 271.1 [192.2 to 382.5] | 180.9 [104.5 to 313.0] | 209.6 [132.1 to 332.5] | 415.7 [298.9 to 578.1] | 68.9 [38.3 to 124.0]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 216.8 [139.0 to 338.1] | 185.0 [104.3 to 328.3] | 226.6 [152.7 to 336.4] | 373.6 [266.6 to 523.6] | 70.4 [42.8 to 115.8]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 126.5 [65.0 to 246.0] |  | 116.1 [58.8 to 229.1] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 413.6 [221.2 to 773.4] |  | 217.4 [99.4 to 475.1] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 384.4 [250.5 to 589.8] |  | 251.7 [150.7 to 420.3] |  |

14. Secondary Outcome: ELISPOT (IFN-g, Peptide Pool: G(B)) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool G(B). Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 111.3 [64.6 to 191.7] | 63.4 [35.4 to 113.3] | 56.8 [31.5 to 102.6] | 135.5 [83.2 to 220.7] | 73.6 [43.6 to 124.1]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 399.6 [243.4 to 656.1] | 306.0 [165.9 to 564.4] | 305.6 [165.5 to 564.2] | 613.0 [428.7 to 876.5] | 65.6 [40.4 to 106.6]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 247.9 [136.5 to 450.1] | 141.4 [73.9 to 270.7] | 181.2 [93.2 to 352.4] | 371.5 [269.7 to 511.7] | 71.6 [43.8 to 117.2]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 196.9 [115.3 to 336.2] | 184.0 [102.6 to 330.0] | 138.8 [73.7 to 261.6] | 406.8 [287.9 to 574.9] | 86.6 [47.4 to 158.3]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 177.8 [102.9 to 307.0] | 219.0 [114.2 to 419.8] | 128.1 [66.4 to 247.3] | 359.7 [257.9 to 501.5] | 77.0 [43.2 to 137.5]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 87.8 [44.5 to 173.3] |  | 57.5 [28.6 to 115.5] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 300.6 [140.3 to 644.0] |  | 101.2 [44.6 to 229.5] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 246.7 [120.0 to 507.3] |  | 132.2 [64.0 to 272.8] |  |

15. Secondary Outcome: ELISPOT (IFN-g, Peptide Pool: M2) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool M2. Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 84.1 [52.2 to 135.6] | 41.2 [29.1 to 58.4] | 54.9 [34.2 to 88.3] | 86.6 [51.4 to 145.9] | 60.5 [38.9 to 94.0]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 353.2 [250.9 to 497.0] | 247.9 [146.6 to 419.0] | 418.8 [245.4 to 714.8] | 352.5 [213.9 to 580.8] | 49.3 [33.0 to 73.9]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 281.9 [197.2 to 403.0] | 136.9 [76.5 to 245.1] | 284.7 [157.1 to 515.7] | 317.9 [217.1 to 465.4] | 42.4 [31.1 to 58.0]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 185.9 [114.8 to 300.8] | 140.5 [80.8 to 244.3] | 208.8 [121.9 to 357.6] | 345.5 [211.2 to 565.2] | 60.4 [36.7 to 99.6]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 208.2 [118.8 to 364.8] | 161.1 [90.9 to 285.6] | 169.6 [94.3 to 305.1] | 333.4 [198.3 to 560.4] | 54.6 [34.2 to 87.2]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 13 | 0 | 0
  Week 56 (Booster Substudy) | 86.8 [44.4 to 169.4] |  | 56.3 [30.2 to 104.9] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 242.0 [126.3 to 463.7] |  | 181.3 [75.9 to 433.1] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 237.0 [122.5 to 458.5] |  | 216.5 [101.0 to 464.2] |  |

16. Secondary Outcome: ELISPOT (IFN-g, Peptide Pool: N) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool N. Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 179.2 [114.8 to 279.7] | 97.1 [62.7 to 150.3] | 85.1 [53.1 to 136.3] | 169.4 [107.9 to 266.2] | 82.7 [51.4 to 132.8]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 652.1 [495.6 to 857.9] | 534.9 [355.4 to 805.1] | 825.9 [591.6 to 1153.0] | 624.2 [421.5 to 924.5] | 86.8 [58.3 to 129.3]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 567.7 [416.2 to 774.4] | 377.2 [223.3 to 637.2] | 521.3 [363.9 to 746.7] | 523.4 [377.4 to 726.0] | 86.5 [57.3 to 130.4]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 452.8 [353.8 to 579.6] | 407.7 [259.4 to 640.9] | 399.7 [292.9 to 545.6] | 513.4 [359.4 to 733.4] | 93.7 [58.0 to 151.3]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 401.3 [306.8 to 524.9] | 401.8 [229.4 to 704.0] | 386.5 [255.7 to 584.0] | 544.0 [401.7 to 736.7] | 78.1 [48.9 to 124.9]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 164.3 [88.4 to 305.6] |  | 166.2 [92.6 to 298.2] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 475.6 [260.9 to 866.8] |  | 385.4 [230.1 to 645.6] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 471.1 [325.7 to 681.4] |  | 436.6 [268.5 to 710.0] |  |

17. Secondary Outcome: ELISPOT (IL-4, Peptide Pool: F) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool F. Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 33.5 [25.0 to 44.9] | 29.2 [24.1 to 35.3] | 44.3 [28.5 to 68.7] | 49.6 [33.8 to 72.6] | 25.0 [25.0 to 25.0]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 28.0 [23.8 to 32.9] | 29.0 [24.4 to 34.4] | 34.1 [24.8 to 46.8] | 34.8 [25.7 to 47.2] | 25.0 [25.0 to 25.0]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 32.8 [24.9 to 43.2] | 35.5 [27.9 to 45.2] | 25.0 [25.0 to 25.0]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 26.6 [23.3 to 30.4] | 25.0 [25.0 to 25.0] | 30.6 [23.9 to 39.2] | 29.1 [24.0 to 35.4] | 25.0 [25.0 to 25.0]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 26.7 [23.2 to 30.7] |  | 26.5 [23.3 to 30.1] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 34.7 [23.6 to 51.1] |  | 28.5 [21.5 to 37.7] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 27.4 [22.5 to 33.4] |  | 27.9 [23.8 to 32.7] |  |

18. Secondary Outcome: ELISPOT (IL-4, Peptide Pool: G(A)) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool G(A). Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 32.0 [23.7 to 43.1] | 27.7 [23.8 to 32.2] | 33.7 [23.2 to 49.0] | 48.2 [33.5 to 69.5] | 25.0 [25.0 to 25.0]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 30.4 [23.9 to 38.7] | 26.6 [23.4 to 30.2] | 31.5 [24.8 to 40.0] | 31.1 [25.0 to 38.7] | 25.0 [25.0 to 25.0]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 26.0 [23.9 to 28.3] | 26.5 [23.5 to 29.8] | 26.0 [24.0 to 28.1] | 33.4 [25.1 to 44.4] | 25.0 [25.0 to 25.0]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 27.3 [22.7 to 32.9] | 31.4 [24.8 to 39.8] | 25.0 [25.0 to 25.0]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 25.0 [25.0 to 25.0] |  | 25.0 [25.0 to 25.0] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 40.4 [23.0 to 70.9] |  | 25.0 [25.0 to 25.0] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 33.0 [23.4 to 46.5] |  | 25.0 [25.0 to 25.0] |  |

19. Secondary Outcome: ELISPOT (IL-4, Peptide Pool: G(B)) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool G(B). Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 30.1 [22.9 to 39.5] | 27.4 [23.9 to 31.5] | 34.2 [23.3 to 50.2] | 43.4 [31.0 to 60.6] | 25.0 [25.0 to 25.0]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 28.1 [21.9 to 36.1] | 27.9 [23.8 to 32.7] | 29.1 [22.9 to 36.8] | 29.5 [24.3 to 35.7] | 25.0 [25.0 to 25.0]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 26.4 [23.5 to 29.7] | 25.0 [25.0 to 25.0] | 26.9 [23.1 to 31.3] | 32.8 [25.8 to 41.7] | 25.0 [25.0 to 25.0]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 27.2 [22.7 to 32.6] | 31.3 [25.0 to 39.3] | 25.0 [25.0 to 25.0]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 26.2 [23.7 to 28.9] |  | 25.0 [25.0 to 25.0] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 38.1 [23.2 to 62.4] |  | 25.0 [25.0 to 25.0] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 29.8 [23.1 to 38.4] |  | 25.0 [25.0 to 25.0] |  |

20. Secondary Outcome: ELISPOT (IL-4, Peptide Pool: M2) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool M2. Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 28.1 [23.8 to 33.2] | 25.9 [24.1 to 27.8] | 39.1 [26.3 to 58.0] | 28.8 [24.3 to 34.1] | 25.0 [25.0 to 25.0]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 28.0 [23.6 to 33.3] | 26.7 [23.2 to 30.7] | 30.8 [22.3 to 42.7] | 27.0 [24.1 to 30.4] | 25.0 [25.0 to 25.0]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 25.0 [25.0 to 25.0] | 26.0 [24.0 to 28.1] | 30.6 [23.6 to 39.6] | 30.0 [24.2 to 37.1] | 25.0 [25.0 to 25.0]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 27.4 [24.0 to 31.2] | 25.0 [25.0 to 25.0] | 28.1 [22.0 to 36.0] | 29.5 [23.2 to 37.4] | 25.0 [25.0 to 25.0]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 25.0 [25.0 to 25.0] |  | 25.0 [25.0 to 25.0] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 28.9 [21.2 to 39.4] |  | 28.1 [21.8 to 36.3] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 26.6 [23.2 to 30.5] |  | 26.7 [23.2 to 30.7] |  |

21. Secondary Outcome: ELISPOT (IL-4, Peptide Pool: N) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool N. Values below the detection limit (DL) are included with a value of '25' (i.e. 1/2 DL)
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study) | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0] | 25.0 [25.0 to 25.0]
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 28.7 [22.9 to 36.0] | 32.9 [25.9 to 41.7] | 41.4 [30.8 to 55.5] | 35.3 [26.1 to 47.9] | 25.0 [25.0 to 25.0]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 26.5 [23.5 to 29.8] | 29.1 [23.4 to 36.3] | 27.9 [23.8 to 32.7] | 30.2 [23.7 to 38.4] | 25.0 [25.0 to 25.0]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 25.0 [25.0 to 25.0] | 30.1 [23.9 to 37.9] | 25.0 [25.0 to 25.0] | 28.0 [23.7 to 33.0] | 25.0 [25.0 to 25.0]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 25.0 [25.0 to 25.0] | 31.3 [24.2 to 40.5] | 27.3 [24.0 to 31.1] | 28.1 [23.6 to 33.5] | 25.0 [25.0 to 25.0]
  Week 56 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 56 (Booster Substudy) | 25.0 [25.0 to 25.0] |  | 25.0 [25.0 to 25.0] |  |
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 28.9 [21.1 to 39.6] |  | 25.0 [25.0 to 25.0] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 27.3 [22.6 to 33.1] |  | 25.0 [25.0 to 25.0] |  |

22. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IFN-g, Peptide Pool: F)
Description: Response rate based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool F. Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 57.1 [34.0 to 78.2] | 95.2 [76.2 to 99.9] | 100.0 [83.2 to 100.0] | 73.9 [51.6 to 89.8] | 8.3 [1.0 to 27.0]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 61.1 [35.7 to 82.7] | 70.0 [45.7 to 88.1] | 95.0 [75.1 to 99.9] | 56.5 [34.5 to 76.8] | 19.0 [5.4 to 41.9]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 23.8 [8.2 to 47.2] | 63.2 [38.4 to 83.7] | 65.0 [40.8 to 84.6] | 56.5 [34.5 to 76.8] | 20.0 [5.7 to 43.7]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 41.2 [18.4 to 67.1] | 61.1 [35.7 to 82.7] | 68.4 [43.4 to 87.4] | 63.6 [40.7 to 82.8] | 10.0 [1.2 to 31.7]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 53.3 [26.6 to 78.7] |  | 21.4 [4.7 to 50.8] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 40.0 [16.3 to 67.7] |  | 14.3 [1.8 to 42.8] |  |

23. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IFN-g, Peptide Pool: G(A))
Description: Response rate based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool G(A). Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 81.0 [58.1 to 94.6] | 81.0 [58.1 to 94.6] | 95.0 [75.1 to 99.9] | 82.6 [61.2 to 95.0] | 8.3 [1.0 to 27.0]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 72.2 [46.5 to 90.3] | 65.0 [40.8 to 84.6] | 85.0 [62.1 to 96.8] | 69.6 [47.1 to 86.8] | 9.5 [1.2 to 30.4]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 38.1 [18.1 to 61.6] | 68.4 [43.4 to 87.4] | 70.0 [45.7 to 88.1] | 65.2 [42.7 to 83.6] | 5.0 [0.1 to 24.9]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 58.8 [32.9 to 81.6] | 66.7 [41.0 to 86.7] | 68.4 [43.4 to 87.4] | 63.6 [40.7 to 82.8] | 5.0 [0.1 to 24.9]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 60.0 [32.3 to 83.7] |  | 50.0 [23.0 to 77.0] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 60.0 [32.3 to 83.7] |  | 57.1 [28.9 to 82.3] |  |

24. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IFN-g, Peptide Pool: G(B))
Description: Response rate based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool G(B). Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 71.4 [47.8 to 88.7] | 76.2 [52.8 to 91.8] | 85.0 [62.1 to 96.8] | 78.3 [56.3 to 92.5] | 12.5 [2.7 to 32.4]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 55.6 [30.8 to 78.5] | 55.0 [31.5 to 76.9] | 70.0 [45.7 to 88.1] | 60.9 [38.5 to 80.3] | 14.3 [3.0 to 36.3]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 42.9 [21.8 to 66.0] | 63.2 [38.4 to 83.7] | 60.0 [36.1 to 80.9] | 65.2 [42.7 to 83.6] | 10.0 [1.2 to 31.7]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 35.3 [14.2 to 61.7] | 61.1 [35.7 to 82.7] | 42.1 [20.3 to 66.5] | 68.2 [45.1 to 86.1] | 5.0 [0.1 to 24.9]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 60.0 [32.3 to 83.7] |  | 57.1 [28.9 to 82.3] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 60.0 [32.3 to 83.7] |  | 42.9 [17.7 to 71.1] |  |

25. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IFN-g, Peptide Pool: M2)
Description: Response rate based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool M2. Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 81.0 [58.1 to 94.6] | 71.4 [47.8 to 88.7] | 95.0 [75.1 to 99.9] | 87.0 [66.4 to 97.2] | 8.3 [1.0 to 27.0]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 72.2 [46.5 to 90.3] | 65.0 [40.8 to 84.6] | 90.0 [68.3 to 98.8] | 65.2 [42.7 to 83.6] | 9.5 [1.2 to 30.4]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 57.1 [34.0 to 78.2] | 78.9 [54.4 to 93.9] | 85.0 [62.1 to 96.8] | 78.3 [56.3 to 92.5] | 15.0 [3.2 to 37.9]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 58.8 [32.9 to 81.6] | 66.7 [41.0 to 86.7] | 68.4 [43.4 to 87.4] | 72.7 [49.8 to 89.3] | 0.0 [0.0 to 16.8]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 13 | 0 | 0
  Week 57 (Booster Substudy) | 66.7 [38.4 to 88.2] |  | 76.9 [46.2 to 95.0] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 13 | 0 | 0
  Week 58 (Booster Substudy) | 60.0 [32.3 to 83.7] |  | 76.9 [46.2 to 95.0] |  |

26. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IFN-g, Peptide Pool: N)
Description: Response rate based on RSV-specific Interferon-gamma (IFN-g) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool N. Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 76.2 [52.8 to 91.8] | 85.7 [63.7 to 97.0] | 100.0 [83.2 to 100.0] | 78.3 [56.3 to 92.5] | 16.7 [4.7 to 37.4]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 72.2 [46.5 to 90.3] | 75.0 [50.9 to 91.3] | 95.0 [75.1 to 99.9] | 60.9 [38.5 to 80.3] | 19.0 [5.4 to 41.9]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 57.1 [34.0 to 78.2] | 84.2 [60.4 to 96.6] | 95.0 [75.1 to 99.9] | 65.2 [42.7 to 83.6] | 20.0 [5.7 to 43.7]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 64.7 [38.3 to 85.8] | 72.2 [46.5 to 90.3] | 73.7 [48.8 to 90.9] | 72.7 [49.8 to 89.3] | 15.0 [3.2 to 37.9]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 60.0 [32.3 to 83.7] |  | 78.6 [49.2 to 95.3] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 80.0 [51.9 to 95.7] |  | 64.3 [35.1 to 87.2] |  |

27. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IL-4, Peptide Pool: F)
Description: Response rate based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool F. Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 19.0 [5.4 to 41.9] | 14.3 [3.0 to 36.3] | 30.0 [11.9 to 54.3] | 47.8 [26.8 to 69.4] | 0.0 [0.0 to 14.2]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 11.1 [1.4 to 34.7] | 15.0 [3.2 to 37.9] | 20.0 [5.7 to 43.7] | 21.7 [7.5 to 43.7] | 0.0 [0.0 to 16.1]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 17.6] | 20.0 [5.7 to 43.7] | 34.8 [16.4 to 57.3] | 0.0 [0.0 to 16.8]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 5.9 [0.1 to 28.7] | 0.0 [0.0 to 18.5] | 15.8 [3.4 to 39.6] | 13.6 [2.9 to 34.9] | 0.0 [0.0 to 16.8]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 20.0 [4.3 to 48.1] |  | 7.1 [0.2 to 33.9] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 6.7 [0.2 to 31.9] |  | 7.1 [0.2 to 33.9] |  |

28. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IL-4, Peptide Pool: G(A))
Description: Response rate based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool G(A). Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 14.3 [3.0 to 36.3] | 9.5 [1.2 to 30.4] | 15.0 [3.2 to 37.9] | 43.5 [23.2 to 65.5] | 0.0 [0.0 to 14.2]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 16.7 [3.6 to 41.4] | 5.0 [0.1 to 24.9] | 20.0 [5.7 to 43.7] | 17.4 [5.0 to 38.8] | 0.0 [0.0 to 16.1]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 4.8 [0.1 to 23.8] | 5.3 [0.1 to 26.0] | 5.0 [0.1 to 24.9] | 17.4 [5.0 to 38.8] | 0.0 [0.0 to 16.8]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5] | 5.3 [0.1 to 26.0] | 18.2 [5.2 to 40.3] | 0.0 [0.0 to 16.8]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 20.0 [4.3 to 48.1] |  | 0.0 [0.0 to 23.2] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 20.0 [4.3 to 48.1] |  | 0.0 [0.0 to 23.2] |  |

29. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IL-4, Peptide Pool: G(B))
Description: Response rate based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool G(B). Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 9.5 [1.2 to 30.4] | 9.5 [1.2 to 30.4] | 15.0 [3.2 to 37.9] | 39.1 [19.7 to 61.5] | 0.0 [0.0 to 14.2]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 5.6 [0.1 to 27.3] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 13.0 [2.8 to 33.6] | 0.0 [0.0 to 16.1]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 4.8 [0.1 to 23.8] | 0.0 [0.0 to 17.6] | 5.0 [0.1 to 24.9] | 21.7 [7.5 to 43.7] | 0.0 [0.0 to 16.8]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5] | 5.3 [0.1 to 26.0] | 18.2 [5.2 to 40.3] | 0.0 [0.0 to 16.8]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 20.0 [4.3 to 48.1] |  | 0.0 [0.0 to 23.2] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 13.3 [1.7 to 40.5] |  | 0.0 [0.0 to 23.2] |  |

30. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IL-4, Peptide Pool: M2)
Description: Response rate based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool M2. Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 9.5 [1.2 to 30.4] | 4.8 [0.1 to 23.8] | 25.0 [8.7 to 49.1] | 13.0 [2.8 to 33.6] | 0.0 [0.0 to 14.2]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 11.1 [1.4 to 34.7] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 8.7 [1.1 to 28.0] | 0.0 [0.0 to 16.1]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 0.0 [0.0 to 16.1] | 5.3 [0.1 to 26.0] | 15.0 [3.2 to 37.9] | 13.0 [2.8 to 33.6] | 0.0 [0.0 to 16.8]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 18.5] | 5.3 [0.1 to 26.0] | 9.1 [1.1 to 29.2] | 0.0 [0.0 to 16.8]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 6.7 [0.2 to 31.9] |  | 7.1 [0.2 to 33.9] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 6.7 [0.2 to 31.9] |  | 7.1 [0.2 to 33.9] |  |

31. Secondary Outcome: Percentage of Participants With Response by ELISPOT (IL-4, Peptide Pool: N)
Description: Response rate based on RSV-specific Interleukin 4 (IL-4) Enzyme-linked Immuno Spot Technique (ELISPOT) for the Peptide Pool N. Response is defined as the appearance of spot forming units ≥ detection limit (50) for initially negative subjects, or a doubling or more of the spot forming units compared to Baseline for initially positive subjects. Response for main study visits is based on main study Baseline, whereas response for booster study visits is based on booster substudy Baseline. Percentages based on number of subjects with paired data available, i.e. number of subjects with results available for the respective time point and the corresponding Baseline.
Time Frame: within 58 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 23 | 24
percentage of subjects
  Week 1 (Main Study): number analyzed (Participants) | 21 | 21 | 20 | 23 | 24
  Week 1 (Main Study) | 9.5 [1.2 to 30.4] | 23.8 [8.2 to 47.2] | 45.0 [23.1 to 68.5] | 21.7 [7.5 to 43.7] | 0.0 [0.0 to 14.2]
  Week 2 (Main Study): number analyzed (Participants) | 18 | 20 | 20 | 23 | 21
  Week 2 (Main Study) | 5.6 [0.1 to 27.3] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 13.0 [2.8 to 33.6] | 0.0 [0.0 to 16.1]
  Week 5 (Main Study): number analyzed (Participants) | 21 | 19 | 20 | 23 | 20
  Week 5 (Main Study) | 0.0 [0.0 to 16.1] | 15.8 [3.4 to 39.6] | 0.0 [0.0 to 16.8] | 8.7 [1.1 to 28.0] | 0.0 [0.0 to 16.8]
  Week 6 (Main Study): number analyzed (Participants) | 17 | 18 | 19 | 22 | 20
  Week 6 (Main Study) | 0.0 [0.0 to 19.5] | 16.7 [3.6 to 41.4] | 10.5 [1.3 to 33.1] | 9.1 [1.1 to 29.2] | 0.0 [0.0 to 16.8]
  Week 57 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 57 (Booster Substudy) | 6.7 [0.2 to 31.9] |  | 0.0 [0.0 to 23.2] |  |
  Week 58 (Booster Substudy): number analyzed (Participants) | 15 | 0 | 14 | 0 | 0
  Week 58 (Booster Substudy) | 6.7 [0.2 to 31.9] |  | 0.0 [0.0 to 23.2] |  |

32. Secondary Outcome: Memory B Cells (IgG) GMSFU
Description: Geometric Mean Spot Forming Units (GMSFUs) based on RSV-specific Immunoglobulin G (IgG)-producing memory B cells. Negative results (i.e. results below 0.01) are included with a value of '0.005'
Time Frame: within 82 weeks
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 13 | 16 | 15 | 18 | 17
Spot Forming Units / 10^6 PBMC
  Week 0 (Main Study): number analyzed (Participants) | 12 | 16 | 15 | 18 | 17
  Week 0 (Main Study) | 0.091 [0.051 to 0.163] | 0.083 [0.046 to 0.151] | 0.068 [0.034 to 0.134] | 0.129 [0.073 to 0.228] | 0.117 [0.061 to 0.225]
  Week 16 (Follow-Up 1): number analyzed (Participants) | 13 | 16 | 14 | 18 | 17
  Week 16 (Follow-Up 1) | 0.171 [0.116 to 0.251] | 0.099 [0.047 to 0.210] | 0.173 [0.087 to 0.344] | 0.210 [0.110 to 0.399] | 0.130 [0.067 to 0.252]
  Week 30 (Follow-Up 2): number analyzed (Participants) | 13 | 16 | 14 | 18 | 17
  Week 30 (Follow-Up 2) | 0.148 [0.093 to 0.237] | 0.068 [0.034 to 0.137] | 0.123 [0.051 to 0.297] | 0.100 [0.053 to 0.189] | 0.079 [0.042 to 0.148]
  Week 56 (Booster Substudy): number analyzed (Participants) | 12 | 0 | 12 | 0 | 0
  Week 56 (Booster Substudy) | 0.127 [0.066 to 0.245] |  | 0.138 [0.072 to 0.266] |  |
  Week 68 (Booster Follow-Up 1): number analyzed (Participants) | 11 | 0 | 13 | 0 | 0
  Week 68 (Booster Follow-Up 1) | 0.104 [0.041 to 0.265] |  | 0.231 [0.111 to 0.480] |  |
  Week 82 (Booster Follow-Up 2): number analyzed (Participants) | 12 | 0 | 11 | 0 | 0
  Week 82 (Booster Follow-Up 2) | 0.103 [0.053 to 0.202] |  | 0.167 [0.088 to 0.318] |  |

33. Secondary Outcome: Serious Adverse Events
Description: Number of participants reporting Serious Adverse Events per period: Between 1st and 2nd vaccination (Vaccination Period 1, Main Study, duration: 4 weeks), between 2nd vaccination and end of active phase of the Main Study (Vaccination Period 2, Main Study, duration: 4 weeks), during the follow-up phase of the Main Study (Follow-Up, Main Study, duration: 22 weeks), after the Main Study and before the booster vaccination (Between Study Parts [retrospectively collected in booster substudy], duration: 26 weeks), between booster vaccination and end of active phase of the Booster Substudy (Booster Vaccination Period, Booster Substudy, duration: 4 weeks), and during the follow-up phase of the Booster Substudy (Follow-Up, Booster Substudy, duration: 48 weeks). Percentages based on number of subjects still in the study at the start of the respective period.
Time Frame: within 108 weeks (Main Study + Booster Substudy)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Vaccination Period 1, Main Study | 0 | 1 | 2 | 1 | 0
  Vaccination Period 2, Main Study: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Vaccination Period 2, Main Study | 1 | 0 | 1 | 0 | 2
  Follow-Up, Main Study: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Follow-Up, Main Study | 1 | 3 | 0 | 1 | 3
  Between Study Parts: number analyzed (Participants) | 44 | 0 | 51 | 0 | 0
  Between Study Parts | 1 |  | 1 |  |
  Booster Vaccination Period, Booster Substudy: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Booster Vaccination Period, Booster Substudy | 0 |  | 0 |  |
  Follow-Up, Booster Substudy: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Follow-Up, Booster Substudy | 1 |  | 0 |  |

34. Secondary Outcome: Related Serious Adverse Events
Description: Number of participants reporting Serious Adverse Events possibly, probably or definitely related to the trial vaccine per period: Between 1st and 2nd vaccination (Vaccination Period 1, Main Study, duration: 4 weeks), between 2nd vaccination and end of active phase of the Main Study (Vaccination Period 2, Main Study, duration: 4 weeks), during the follow-up phase of the Main Study (Follow-Up, Main Study, duration: 22 weeks), after the Main Study and before the booster vaccination (Between Study Parts [retrospectively collected in booster substudy], duration: 26 weeks), between booster vaccination and end of active phase of the Booster Substudy (Booster Vaccination Period, Booster Substudy, duration: 4 weeks), and during the follow-up phase of the Booster Substudy (Follow-Up, Booster Substudy, duration: 48 weeks). Percentages based on number of subjects still in the study at the start of the respective period.
Time Frame: within 108 weeks (Main Study + Booster Substudy)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Vaccination Period 1, Main Study | 0 | 0 | 0 | 0 | 0
  Vaccination Period 2, Main Study: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Vaccination Period 2, Main Study | 0 | 0 | 0 | 0 | 0
  Follow-Up, Main Study: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Follow-Up, Main Study | 0 | 0 | 0 | 0 | 0
  Between Study Parts: number analyzed (Participants) | 44 | 0 | 51 | 0 | 0
  Between Study Parts | 0 |  | 0 |  |
  Booster Vaccination Period, Booster Substudy: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Booster Vaccination Period, Booster Substudy | 0 | 0 | 0 | 0 | 0
  Follow-Up, Booster Substudy: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Follow-Up, Booster Substudy | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Grade ≥ 3 Serious Adverse Events
Description: Number of participants reporting Serious Adverse Events with intensity ≥ Grade 3 per period: Between 1st and 2nd vaccination (Vaccination Period 1, Main Study, duration: 4 weeks), between 2nd vaccination and end of active phase of the Main Study (Vaccination Period 2, Main Study, duration: 4 weeks), during the follow-up phase of the Main Study (Follow-Up, Main Study, duration: 22 weeks), after the Main Study and before the booster vaccination (Between Study Parts [retrospectively collected in booster substudy], duration: 26 weeks), between booster vaccination and end of active phase of the Booster Substudy (Booster Vaccination Period, Booster Substudy, duration: 4 weeks), and during the follow-up phase of the Booster Substudy (Follow-Up, Booster Substudy, duration: 48 weeks). Percentages based on number of subjects still in the study at the start of the respective period.
Time Frame: within 108 weeks (Main Study + Booster Substudy)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Vaccination Period 1, Main Study | 0 | 1 | 1 | 1 | 0
  Vaccination Period 2, Main Study: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Vaccination Period 2, Main Study | 1 | 0 | 1 | 0 | 1
  Follow-Up, Main Study: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Follow-Up, Main Study | 1 | 3 | 0 | 0 | 2
  Between Study Parts: number analyzed (Participants) | 44 | 0 | 51 | 0 | 0
  Between Study Parts | 1 |  | 1 |  |
  Booster Vaccination Period, Booster Substudy: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Booster Vaccination Period, Booster Substudy | 0 |  | 0 |  |
  Follow-Up, Booster Substudy: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Follow-Up, Booster Substudy | 1 |  | 0 |  |

36. Secondary Outcome: Related Grade ≥ 3 Adverse Events
Description: Number of participants reporting Adverse Events possibly, probably or definitely related to the trial vaccine with intensity ≥ Grade 3 per period: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Pooled solicited (general only) and unsolicited AEs. Percentages based on number of subjects still in the study at the start of the respective period.
Time Frame: within 29 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Vaccination Period 1, Main Study | 0 | 3 | 6 | 6 | 0
  Vaccination Period 2, Main Study: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Vaccination Period 2, Main Study | 3 | 1 | 1 | 2 | 0
  Booster Vaccination Period, Booster Substudy: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Booster Vaccination Period, Booster Substudy | 3 |  | 2 |  |

37. Secondary Outcome: Solicited Local Adverse Events
Description: Incidence of injection site reactions (solicited via diary cards) after vaccination: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Percentages based on number of subjects with a completed diary card for the respective vaccination period.
Time Frame: within 8 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Pain - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Pain - Vaccination Period 1 | 39 | 57 | 58 | 76 | 9
  Pain - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Pain - Vaccination Period 2 | 6 | 39 | 6 | 51 | 10
  Pain - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Pain - Booster Vaccination Period | 24 |  | 39 |  |
  Erythema - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Erythema - Vaccination Period 1 | 15 | 13 | 24 | 19 | 14
  Erythema - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Erythema - Vaccination Period 2 | 5 | 13 | 6 | 17 | 8
  Erythema - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Erythema - Booster Vaccination Period | 9 |  | 15 |  |
  Swelling - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Swelling - Vaccination Period 1 | 11 | 13 | 16 | 17 | 2
  Swelling - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Swelling - Vaccination Period 2 | 1 | 8 | 1 | 16 | 1
  Swelling - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Swelling - Booster Vaccination Period | 9 |  | 15 |  |
  Induration - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Induration - Vaccination Period 1 | 9 | 5 | 13 | 13 | 3
  Induration - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Induration - Vaccination Period 2 | 0 | 2 | 3 | 11 | 3
  Induration - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Induration - Booster Vaccination Period | 7 |  | 13 |  |
  Pruritis - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Pruritis - Vaccination Period 1 | 3 | 7 | 14 | 7 | 4
  Pruritis - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Pruritis - Vaccination Period 2 | 2 | 10 | 2 | 5 | 1
  Pruritis - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Pruritis - Booster Vaccination Period | 3 |  | 11 |  |

38. Secondary Outcome: Grade ≥ 3 Solicited Local Adverse Events
Description: Incidence of injection site reactions (solicited via diary cards) with intensity ≥ Grade 3 after vaccination: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Percentages based on number of subjects with a completed diary card for the respective vaccination period.
Time Frame: within 8 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Grade ≥ 3 Pain - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Pain - Vaccination Period 1 | 0 | 0 | 2 | 7 | 0
  Grade ≥ 3 Pain - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Pain - Vaccination Period 2 | 0 | 0 | 1 | 1 | 0
  Grade ≥ 3 Pain - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Pain - Booster Vaccination Period | 2 |  | 4 |  |
  Grade ≥ 3 Erythema - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Erythema - Vaccination Period 1 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Erythema - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Erythema - Vaccination Period 2 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Erythema - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Erythema - Booster Vaccination Period | 0 |  | 0 |  |
  Grade ≥ 3 Swelling - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Swelling - Vaccination Period 1 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Swelling - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Swelling - Vaccination Period 2 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Swelling - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Swelling - Booster Vaccination Period | 0 |  | 0 |  |
  Grade ≥ 3 Induration - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Induration - Vaccination Period 1 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Induration - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Induration - Vaccination Period 2 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Induration - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Induration - Booster Vaccination Period | 0 |  | 0 |  |
  Grade ≥ 3 Pruritis - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Pruritis - Vaccination Period 1 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Pruritis - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Pruritis - Vaccination Period 2 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Pruritis - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Pruritis - Booster Vaccination Period | 0 |  | 1 |  |

39. Secondary Outcome: Solicited General Adverse Events
Description: Incidence of systemic reactions (solicited via diary cards) after vaccination: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Percentages based on number of subjects with a completed diary card for the respective vaccination period.
Time Frame: within 8 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Fever - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Fever - Vaccination Period 1 | 2 | 4 | 8 | 6 | 1
  Fever - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Fever - Vaccination Period 2 | 0 | 0 | 2 | 0 | 0
  Fever - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Fever - Booster Vaccination Period | 0 |  | 3 |  |
  Headache - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Headache - Vaccination Period 1 | 4 | 16 | 21 | 21 | 13
  Headache - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Headache - Vaccination Period 2 | 7 | 14 | 8 | 16 | 9
  Headache - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Headache - Booster Vaccination Period | 9 |  | 13 |  |
  Myalgia - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Myalgia - Vaccination Period 1 | 13 | 19 | 37 | 34 | 7
  Myalgia - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Myalgia - Vaccination Period 2 | 5 | 14 | 5 | 21 | 8
  Myalgia - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Myalgia - Booster Vaccination Period | 10 |  | 24 |  |
  Chills - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Chills - Vaccination Period 1 | 5 | 4 | 10 | 11 | 3
  Chills - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Chills - Vaccination Period 2 | 3 | 2 | 5 | 10 | 7
  Chills - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Chills - Booster Vaccination Period | 3 |  | 4 |  |
  Nausea - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Nausea - Vaccination Period 1 | 2 | 6 | 4 | 6 | 4
  Nausea - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Nausea - Vaccination Period 2 | 7 | 3 | 2 | 6 | 1
  Nausea - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Nausea - Booster Vaccination Period | 1 |  | 3 |  |
  Fatigue - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Fatigue - Vaccination Period 1 | 7 | 15 | 22 | 26 | 5
  Fatigue - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Fatigue - Vaccination Period 2 | 8 | 9 | 4 | 15 | 10
  Fatigue - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Fatigue - Booster Vaccination Period | 4 |  | 16 |  |

40. Secondary Outcome: Grade ≥ 3 Solicited General Adverse Events
Description: Incidence of systemic reactions (solicited via diary cards) with intensity ≥ Grade 3 after vaccination: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Percentages based on number of subjects with a completed diary card for the respective vaccination period.
Time Frame: within 8 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Grade ≥ 3 Fever - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Fever - Vaccination Period 1 | 0 | 1 | 0 | 0 | 0
  Grade ≥ 3 Fever - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Fever - Vaccination Period 2 | 0 | 0 | 0 | 0 | 0
  Grade ≥ 3 Fever - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Fever - Booster Vaccination Period | 0 |  | 0 |  |
  Grade ≥ 3 Headache - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Headache - Vaccination Period 1 | 0 | 1 | 2 | 0 | 1
  Grade ≥ 3 Headache - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Headache - Vaccination Period 2 | 1 | 1 | 0 | 0 | 0
  Grade ≥ 3 Headache - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Headache - Booster Vaccination Period | 2 |  | 0 |  |
  Grade ≥ 3 Myalgia - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Myalgia - Vaccination Period 1 | 0 | 1 | 4 | 3 | 0
  Grade ≥ 3 Myalgia - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Myalgia - Vaccination Period 2 | 2 | 1 | 1 | 1 | 0
  Grade ≥ 3 Myalgia - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Myalgia - Booster Vaccination Period | 1 |  | 2 |  |
  Grade ≥ 3 Chills - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Chills - Vaccination Period 1 | 0 | 0 | 3 | 1 | 0
  Grade ≥ 3 Chills - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Chills - Vaccination Period 2 | 1 | 0 | 0 | 1 | 0
  Grade ≥ 3 Chills - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Chills - Booster Vaccination Period | 0 |  | 0 |  |
  Grade ≥ 3 Nausea - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Nausea - Vaccination Period 1 | 0 | 0 | 1 | 0 | 0
  Grade ≥ 3 Nausea - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Nausea - Vaccination Period 2 | 1 | 0 | 0 | 0 | 0
  Grade ≥ 3 Nausea - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Nausea - Booster Vaccination Period | 0 |  | 0 |  |
  Grade ≥ 3 Fatigue - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Grade ≥ 3 Fatigue - Vaccination Period 1 | 0 | 0 | 4 | 2 | 1
  Grade ≥ 3 Fatigue - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Grade ≥ 3 Fatigue - Vaccination Period 2 | 3 | 0 | 1 | 2 | 0
  Grade ≥ 3 Fatigue - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Grade ≥ 3 Fatigue - Booster Vaccination Period | 0 |  | 1 |  |

41. Secondary Outcome: Related Solicited General Adverse Events
Description: Incidence of systemic reactions (solicited via diary cards) possibly, probably or definitely related to the trial vaccine after vaccination: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Percentages based on number of subjects with a completed diary card for the respective vaccination period.
Time Frame: within 8 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Related Fever - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Related Fever - Vaccination Period 1 | 2 | 4 | 7 | 3 | 1
  Related Fever - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Related Fever - Vaccination Period 2 | 0 | 0 | 2 | 0 | 0
  Related Fever - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Related Fever - Booster Vaccination Period | 0 |  | 2 |  |
  Related Headache - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Related Headache - Vaccination Period 1 | 4 | 14 | 15 | 17 | 7
  Related Headache - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Related Headache - Vaccination Period 2 | 5 | 12 | 4 | 12 | 6
  Related Headache - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Related Headache - Booster Vaccination Period | 7 |  | 12 |  |
  Related Myalgia - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Related Myalgia - Vaccination Period 1 | 9 | 18 | 29 | 29 | 6
  Related Myalgia - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Related Myalgia - Vaccination Period 2 | 5 | 12 | 3 | 18 | 6
  Related Myalgia - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Related Myalgia - Booster Vaccination Period | 10 |  | 23 |  |
  Related Chills - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Related Chills - Vaccination Period 1 | 4 | 4 | 8 | 11 | 3
  Related Chills - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Related Chills - Vaccination Period 2 | 3 | 2 | 5 | 8 | 4
  Related Chills - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Related Chills - Booster Vaccination Period | 3 |  | 4 |  |
  Related Nausea - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Related Nausea - Vaccination Period 1 | 1 | 5 | 4 | 5 | 3
  Related Nausea - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Related Nausea - Vaccination Period 2 | 6 | 2 | 2 | 5 | 1
  Related Nausea - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Related Nausea - Booster Vaccination Period | 1 |  | 3 |  |
  Related Fatigue - Vaccination Period 1: number analyzed (Participants) | 78 | 87 | 79 | 90 | 83
  Related Fatigue - Vaccination Period 1 | 7 | 12 | 18 | 23 | 3
  Related Fatigue - Vaccination Period 2: number analyzed (Participants) | 75 | 83 | 78 | 89 | 81
  Related Fatigue - Vaccination Period 2 | 8 | 9 | 4 | 14 | 8
  Related Fatigue - Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Related Fatigue - Booster Vaccination Period | 4 |  | 15 |  |

42. Secondary Outcome: Unsolicited Non-serious Adverse Events
Description: Incidence of unsolicited non-serious adverse events by period: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Percentages based on number of subjects having received the respective vaccination.
Time Frame: within 29 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Vaccination Period 1 | 14 | 23 | 23 | 22 | 21
  Vaccination Period 2: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Vaccination Period 2 | 21 | 23 | 26 | 21 | 27
  Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Booster Vaccination Period | 1 |  | 3 |  |

43. Secondary Outcome: Related Unsolicited Non-serious Adverse Events
Description: Incidence of unsolicited non-serious adverse events possibly, probably or definitely related to the trial vaccine by period: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Percentages based on number of subjects having received the respective vaccination.
Time Frame: within 29 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Vaccination Period 1 | 4 | 6 | 9 | 9 | 4
  Vaccination Period 2: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Vaccination Period 2 | 4 | 2 | 5 | 6 | 9
  Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Booster Vaccination Period | 0 |  | 3 |  |

44. Secondary Outcome: Grade ≥ 3 Unsolicited Non-serious Adverse Events
Description: Incidence of unsolicited non-serious adverse events with intensity ≥ Grade 3 by period: Following the 1st vaccination (Vaccination Period 1, Main Study), following the 2nd vaccination (Vaccination Period 2, Main Study), and following the booster vaccination (Booster Vaccination Period, Booster Substudy). Percentages based on number of subjects having received the respective vaccination.
Time Frame: within 29 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
Number analyzed (Participants) | 78 | 89 | 80 | 90 | 83
Participants
  Vaccination Period 1 | 1 | 0 | 3 | 0 | 0
  Vaccination Period 2: number analyzed (Participants) | 76 | 84 | 78 | 90 | 82
  Vaccination Period 2 | 2 | 0 | 1 | 0 | 2
  Booster Vaccination Period: number analyzed (Participants) | 43 | 0 | 45 | 0 | 0
  Booster Vaccination Period | 0 |  | 0 |  |

ADVERSE EVENTS:
Time Frame: 108 weeks for participants of both study parts and 30 weeks for participants of the main study only
Description: Serious adverse events were to be reported during the entire study, non-serious adverse events within 4 weeks after each vaccination. Percentages of participants are based on MedDRA Preferred Terms.
Arm/Group | Group 1 - Single Low Dose / Booster | Group 2 - Two Low Doses | Group 3 - Single High Dose / Booster | Group 4 - Two High Doses | Group 5 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/89 | 0/80 | 0/90 | 0/83
Serious Adverse Events (participants affected / at risk) | 4/78 | 4/89 | 4/80 | 2/90 | 5/83
Other Adverse Events (participants affected / at risk) | 15/78 | 23/89 | 20/80 | 28/90 | 27/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Single Low Dose / Booster (N=78) | Group 2 - Two Low Doses (N=89) | Group 3 - Single High Dose / Booster (N=80) | Group 4 - Two High Doses (N=90) | Group 5 - Placebo (N=83)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Single Low Dose / Booster (N=78) | Group 2 - Two Low Doses (N=89) | Group 3 - Single High Dose / Booster (N=80) | Group 4 - Two High Doses (N=90) | Group 5 - Placebo (N=83)
Fatigue (General disorders) | 2 | 0 | 4 | 0 | 1
Injection site pain (General disorders) | 1 | 2 | 4 | 5 | 0
Injection site swelling (General disorders) | 1 | 0 | 4 | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 6 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 6 | 5 | 10
Blood sodium increased (Investigations) | 0 | 1 | 1 | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 4 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 4 | 8 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 4 | 6 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 5 | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02873286/SAP_000.pdf
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT02873286/Prot_001.pdf